CLINICAL TRIAL: NCT06931782
Title: Effectiveness of Artificial Intelligence (AI) in the Prevention, Diagnosis, and Triage of Respiratory Diseases: A Multicenter, Randomized Controlled Study
Brief Title: AI in Respiratory Disease Prevention, Diagnosis, and Triage
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Jianxing He, Professor, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AI-RD-PDT-250323-001
Record Dates: First submitted 2025-03-26; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Respiratory Diseases; Artificial Intelligence (AI); Randomized Controlled Trial
MeSH Terms: conditions — Respiratory Tract Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- AI-Assisted Group (Experimental): Participants completed the questionnaire using AI-driven tools for content generation and information retrieval.
  Interventions: Other: AI
- Internet-Based Group (No Intervention): Participants completed the questionnaire using standard internet search engines for information retrieval.

INTERVENTIONS:
Other: AI — GPT-4o fine-tuned with the Lungdiag database
  Arms: AI-Assisted Group

SUMMARY:
This study will evaluate the impact of using the GPT-4o compared to traditional online tools in the field of respiratory disease prevention, focusing on the dissemination of knowledge and behavior changes among the general public. We will explore the effectiveness of GPT-4o in enhancing public awareness and management capabilities regarding respiratory diseases and promoting appropriate preventive behaviors.

DETAILED DESCRIPTION:
Artificial intelligence (AI) technologies, particularly advanced large language models like GPT-4o developed by OpenAI, hold immense potential in enhancing public health education and preventive behaviors. Although GPT-4o was not specifically designed for respiratory disease prevention, it has shown promising prospects in numerous healthcare-related applications, such as providing health information, responding to public inquiries, and supporting health education efforts. However, its effectiveness in improving public awareness and management capabilities regarding respiratory diseases remains to be further explored.

Understanding and managing respiratory diseases involve complex processes, including symptom recognition, application of preventive knowledge, and informed decision-making. Integrating AI tools like GPT-4o into public health education could potentially enhance knowledge dissemination, reduce misinformation, and encourage appropriate preventive behaviors among the general population. Nevertheless, GPT-4o has not been specifically validated for respiratory disease prevention and carries the risk of generating misleading or inaccurate information, which could confuse users. Improper use of such tools may fail to raise awareness and could even lead to counterproductive behaviors. Therefore, studying how large language models like GPT-4o can effectively support public education and behavior change in this context is of critical importance.

In this study, participants will be randomly divided into two groups: one group will have access to Fine-turned GPT-4o, while the other will rely solely on traditional online tools. They will be presented with scenarios related to respiratory diseases and asked to explain their identification of high-risk factors, understanding of diagnoses, and proposed triage actions for each scenario. Each scenario was developed by a panel of three experts in respiratory health, who also established standardized answers. Responses will be evaluated by two independent groups of reviewers unaware of the participants' group assignments. These experts independently created initial scoring criteria and resolved discrepancies through multiple rounds of discussion to ensure consistency and accuracy.

ELIGIBILITY:
Inclusion Criteria:

* No medical background
* Aged from 18 to 75 years old

Exclusion Criteria:

* Had a medical background
* Exceeds the age criteria
* Failed to comply with the survey requirements

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2400 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
the accuracy of participants in answering questions related to triage, diagnosis, and risk factor identification of respiratory diseases using artificial intelligence versus internet-based information retrieval assessed by questionnaire survey | From enrollment to the end of test at 1 hour.

SECONDARY OUTCOMES:
the accuracy of different subgroups in answering questions related to triage, diagnosis, and risk factor identification of respiratory diseases using artificial intelligence versus internet-based information retrieval assessed by questionnaire survey | From enrollment to the end of test at 1 hour.
Time (in seconds) participants spend per questionnaire between the two study arms. | From enrollment to the end of test at 1 hour.

CONTACTS AND LOCATIONS:
Locations (1):
- the First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong 510120, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes
This study aims to evaluate the effectiveness of artificial intelligence (AI) in the prevention, diagnosis, and triage of respiratory diseases, utilizing a multicenter, randomized controlled trial design. A total of 2400 participants aged 18 to 75 without a medical background will be recruited and randomly assigned to two groups: one group will complete surveys with the assistance of AI tools, while the other group will use standard internet resources to fill out the surveys. The primary outcome measures will include triage accuracy rates, preliminary diagnosis compliance rates, and completeness of risk factor identification, while secondary outcomes will focus on variations in performance across different regions and the lifestyle habits and health indicators of participants. To ensure data quality, training will be conducted at each center, with real-time data entry and auditing processes established. The study plan also includes emergency response protocols and data security manage
Supporting Information: Study Protocol